CLINICAL TRIAL: NCT00195871
Title: A Multicenter, Phase 2 Study, to Evaluate Safety and Efficacy of an Acute Lymphoblastic Leukemia (ALL) Intensive Chemotherapy for Adult Lymphoblastic Lymphoma (LL).
Brief Title: Safety and Efficacy of an Adult Acute Lymphoblastic Leukemia Chemotherapy for Adult Lymphoblastic Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Principal Investigator, Stephane Lepretre, Principal Investigator, Centre Henri Becquerel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LL03
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Lymphoblastic Lymphoma
Keywords: Non-Hodgkin; Lymphoma; Lymphoblastic
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma | interventions — Prednisone; Vincristine; Daunorubicin; Cyclophosphamide; Asparaginase; Cytarabine; Methotrexate; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Prednisone, vincristine, daunorubicin , cyclophosphamide , L.-asparaginase, cytosine-arabinoside, methotrexate, etoposide — coventional dosages
  Other Names: nono
Procedure: hematopoietic stem cell allograft — conventional procedures

SUMMARY:
The primary objective of this study is to evaluate the safety and the efficacy of an adult "acute lymphoblastic leukaemia" type chemotherapy in patients less than 60 years with lymphoblastic lymphoma. Treatment principle is based on an intensive induction and a delayed intensification.

DETAILED DESCRIPTION:
Lymphoblastic lymphomas (LL) are rare and represent less than 2% of the malignant non-Hodgkin lymphomas (NHL). The distinction between a LL and an acute lymphoblastic leukaemia (ALL) is difficult; it is arbitrarily based on the percentage of medullary blasts. Above 20% of blasts, it is an ALL. In both cases, the same type of cells is affected: the lymphoblast. Thus the LL were treated either as aggressive NHL or as ALL. The results of the various clinical studies, have shown a best efficacy of ALL type treatments(in terms of overall survival and disease free survival). These treatments are based on an induction phase with reinforced cyclophosphamide and L-asparaginase, and a re-use of the first drugs after consolidation (delayed intensification). The prognostic factors of ALL are now better defined, determining risk groups. According to these prognostic indicators, the allograft could be proposed in first complete remission. Indicators are biological (hyperleukocytosis, chromosomal abnormalities as t(4;11), t(9;22), t(1;19) translocations), clinical (central nervous system involvement), evolutive (salvage therapy needed to obtain complete remission), consideration of early response (cortico-sensibility and chemo-sensibility) and molecular responses (residual disease). On the other hand, the prognostic factors of LL are not well known. This study should permit to better define them. So the prognostic indicators of ALL, in this study, will be decisional for the indication of allograft. This treatment is based on a parallel currently recruiting adult patients with ALL (protocol GRAALL 2003).

ELIGIBILITY:
Inclusion Criteria:

* Patient with lymphoblastic lymphoma.
* Aged from 18 to 59 years.
* Medullary blasts rate less than 20%
* Non previously treated
* With or without central nervous system or meningeal involvement.
* No contra-indication to anthracyclines.
* No contra-indication to intensive treatments
* Negative HIV serology test
* Negative pregnancy test for all female patients of childbearing potential.
* Able to be regularly followed up.

Exclusion Criteria:

* Evolutive cancer with the exception of non melanoma skin tumours or stage 0 (in situ) cervical carcinoma.
* Prior treatment with chemotherapy.
* Lymphoblastic Transformation of chronic myeloid leukaemia
* Patient unable to be regularly followed-up.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2004-02; Primary Completion 2014-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 2 y

SECONDARY OUTCOMES:
Disease Free Survival ; Complete response rate ; Overall Survival ; Progression rate; Relapse rate ; Central Nervous System or meningeal relapse rate ; medullary relapse rate ; toxicities. | 2 y

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Lepretre, MD, Study Chair — Centre Henri Becquerel, Rouen, France; Hervé Dombret, MD, Principal Investigator — Saint-Louis Hospital, Paris, France; Norbert Ifrah, MD, Principal Investigator — Centre Hospitalier Universitaire d'Angers, FRANCE
Locations (19):
- Belgium (2):
  - Chr de La Citadelle, Liège
  - Cliniques Universitaires U C L de Mont Godinne, Yvoir
- France (17):
  - C H U D'Angers, Angers
  - Centre Hospitalier de La Region Annecienne, Annecy
  - Chu de Grenoble, Grenoble
  - Centre Hospitalier de Lens, Lens
  - Edouard Herriot Hospital, Lyon
  - Pierre Benite Hospital, Lyon
  - Institut Paoli Calmettes, Marseille
  - Saint-Louis Hospital, Paris
  - La Pitie Salpetriere Hospital, Paris
  - Cochin Hospital, Paris
  - Marechal Joffre Hospital, Perpignan
  - Centre Hospitalier de Poitiers, Poitiers
  - Chu de Reims Robert Debre Hospital, Reims
  - Centre Henri Becquerel, Rouen
  - Institut de Cancerologie de La Loire, Saint-Priest-en-Jarez
  - Bretonneau Hospital, Tours
  - Chu de Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Le Gouill S, Lepretre S, Briere J, Morel P, Bouabdallah R, Raffoux E, Sebban C, Lepage E, Brice P. Adult lymphoblastic lymphoma: a retrospective analysis of 92 patients under 61 years included in the LNH87/93 trials. Leukemia. 2003 Nov;17(11):2220-4. doi: 10.1038/sj.leu.2403095. PMID 14576732
- See also: Official site of the Groupe d'Etudes des Lymphomes de l'Adulte (In French) — http://www.gela.org